CLINICAL TRIAL: NCT04182815
Title: Transbronchial Biopsy Assisted by Robot Guidance in the Evaluation of Tumors
Brief Title: Transbronchial Biopsy Assisted by Robot Guidance in the Evaluation of Tumors of the Lung
Acronym: TARGET
Status: Completed | Type: Observational
Sponsor: Auris Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 19-BR-0001
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Nodule; Lung Cancer
Keywords: Bronchoscopy; Robotic bronchoscopy; Lung Lesions; Peripheral lesions; Lung Cancer; Monarch
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Robotic assisted bronchoscopy: Robotic assisted bronchoscopy procedures will be performed using the Monarch platform.
  Interventions: Device: Robotic assisted bronchoscopy

INTERVENTIONS:
Device: Robotic assisted bronchoscopy — Robotic assisted bronchoscopy of peripheral airways in human subjects for the purpose of biopsying peripheral lung lesions.
  Other Names: Robotic assisted bronchoscopy with Monarch platform

SUMMARY:
This study is designed to evaluate clinical safety and diagnostic accuracy of the robotic-assisted bronchoscopy with biopsy performed with the Monarch™ Endoscopy Platform in a broad range of patients with pulmonary lesions.

DETAILED DESCRIPTION:
Despite technological advancements in guided bronchoscopy such as electromagnetic navigation bronchoscopy and radial probe endobronchial ultrasound, successful biopsy of peripheral pulmonary lesions remains a challenge due to a number of factors, one of which may be the ability to gain access to peripheral lesions due to the size and maneuverability of conventional bronchoscopes. The diagnostic yield of conventional bronchoscopic approaches for peripheral lesions remains suboptimal.

A novel robotic assisted bronchoscopy procedure now exists for patients with lung nodules. This procedure is performed using the Monarch™ platform (Auris Health, Inc., Redwood City, CA). This study is expected to enroll up to 1200 patients at up to 30 investigative sites.

ELIGIBILITY:
Inclusion Criteria:

1. Over 21 years of age;
2. Capable and willing to give informed consent;
3. Acceptable candidate for an elective, non-emergent bronchoscopic procedure;
4. Lung lesions, 8 mm to 50 mm in size, requiring bronchoscopic diagnosis which were identified on thin slice CT scan within 28 days of the intended bronchoscopy

Exclusion Criteria:

1. Medical contraindication to bronchoscopy as assessed by the investigator
2. Presence of uncorrectable bleeding disorders
3. Medical devices interfering with electro-magnetic navigation, including but not limited to pacemaker
4. Patients with the target lesion having endobronchial involvement seen on chest CT
5. Lack fitness to undergo flexible bronchoscopy as determined by the bronchoscopist prior to procedure,
6. Participation in any other clinical trial within 30 days of enrollment that would interfere with this study;
7. Uncontrolled or irreversible coagulopathy;
8. Female subjects who are pregnant or nursing at the time of the procedure or those of child-bearing potential refusing a pregnancy test prior to the procedure;
9. CT scan done greater than 28 days before the bronchoscopy procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indeterminate pulmonary nodules considered to undergo a bronchoscopy procedure per standard of care.
Sampling Method: Probability Sample
Enrollment: 691 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of device or procedure related complications | up to 7 days post procedure
  The primary endpoint is a composite that includes pneumothorax requiring intervention rated as > Grade 1 according to the Common Terminology Criteria for Adverse Events (CTCAE) scale, bleeding requiring medical intervention, rated as > Grade 1 according to the CTCAE scale, and respiratory failure, rated as > Grade 3 according to the CTCAE scale.

SECONDARY OUTCOMES:
Rate of device or procedure related complications | up to 7 days post procedure
  Individual components of the primary endpoint
Rate of all pneumothoraxes | up to 7 days post procedure
Total procedure time | During the procedure
Rate of conversion to conventional bronchoscopic procedure | During the procedure
Rate of adverse events unrelated to device or procedure | up to 7 days post procedure
Stage at diagnosis | up to 24 months post procedure
  Stage at diagnosis (if applicable) will be evaluated for all robotic-assisted bronchoscopy procedures performed for suspicion of lung cancer
Diagnostic yield | up to 24 months post procedure
  Diagnostic yield for all robotic-assisted procedure performed for suspicion of lung cancer will be evaluated based on histopathological assessment of acquired tissue samples
Sensitivity for malignancy | up to 24 months post procedure
Rate of post-bronchoscopy infections | up to 7 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Septimiu Murgu, MD, Principal Investigator — University of Chicago
Locations (19):
- United States (17):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Costal Pulmonary Associates, Encinitas, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - The University of Connecticut Health Center, Farmington, Connecticut
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Spectrum Health System, Grand Rapids, Michigan
  - Minnesota Lung Center, Ltd, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - University of Pittsburgh Medical Center, Hamot, Erie, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - TriStar Centennial Medical Center, Nashville, Tennessee
- University Health Network, Toronto, Ontario, Canada
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murgu S, Chen AC, Gilbert CR, Sterman DH, Pederson D, Rafeq S, Laxmanan B, Schwiers ML, Connelly J, Benz HL, Yasufuku K, Silvestri GA; TARGET Investigators. A Prospective, Multicenter Evaluation of Safety and Diagnostic Outcomes With Robotic-Assisted Bronchoscopy: Results of the Transbronchial Biopsy Assisted by Robot Guidance in the Evaluation of Tumors of the Lung (TARGET) Trial. Chest. 2025 Aug;168(2):539-555. doi: 10.1016/j.chest.2025.04.022. Epub 2025 Apr 27. PMID 40300665
- [Derived] Agrawal A. Interventional Pulmonology: Diagnostic and Therapeutic Advances in Bronchoscopy. Am J Ther. 2021 Feb 9;28(2):e204-e216. doi: 10.1097/MJT.0000000000001344. PMID 33590989